CLINICAL TRIAL: NCT05023278
Title: The Use of Venlafaxine in Reducing Acute Post-Surgical Pain and Opioid Consumption in Primary Total Knee Replacement
Brief Title: The Use of Venlafaxine in Reducing Pain in Primary Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-32595
Record Dates: First submitted 2021-07-19; First posted 2021-08-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Pain; Chronic Pain; Knee Pain Chronic; Neuropathic Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain; Neuralgia | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects in placebo arm will receive inactive placebo capsule daily for 7 consecutive days starting on day of primary arthroplasty surgery.
  Interventions: Drug: Placebo
- Venlafaxine (Experimental): Subjects in venlafaxine arm will receive venlafaxine 37.5mg daily for 7 consecutive days starting on day of primary arthroplasty surgery.
  Interventions: Drug: Venlafaxine 37.5 MG

INTERVENTIONS:
Drug: Venlafaxine 37.5 MG — venlafaxine 37.5mg daily for 7 consecutive days.
  Other Names: SNRI analgesia
  Arms: Venlafaxine
Drug: Placebo — placebo filled pill daily for 7 consecutive days.
  Other Names: control
  Arms: Placebo

SUMMARY:
Patients experience pain after their knee replacement surgery - and some may continue to experience persistent pain long after their knee replacement surgery. Traditional pain management strategies reply on pain medication such as opioids for pain control. However, these drugs do not work well for pain associated with movement or the the nerve pain (tingling, electrical sensations) after surgery. In addition, opioids are associated with significant side effects such as nausea, vomiting, respiratory depression, depression, cognitive dysfunction and risk of persistent opioid use. Neuropathic pain medications, such as venlafaxine are effective in managing nerve pain. Recent studies also support its potential role in acute pain management. Here, we propose a prospective randomized clinical trial 1) to evaluate the efficacy of Venlafaxine in reducing pain intensity and opioid consumption at post-operative day 1 (POD1) and 1- week after surgery, and 2) to examine whether the use of Venlafaxine will reduce the incidents of chronic postsurgical pain in TKA patients at 3-month time point.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will be randomized to receive either Venlafaxine extended release (ER) 37.5 mg/d or a placebo on the day of surgery and continue the treatment for 7 days after surgery. The primary outcomes include pain severity score (numeric rating scale, NRS) and consumption of morphine miligram equivalent (MME) at 24 hours. The secondary outcome will measure MME and NRS at postoperative day 7. In addition, the disability scale and perceived function 3 months after surgery will be compared to the baseline level by using PROMIS (Patient-Reported Outcomes Measurement Information System)10 Global Health, KOOS, JR. (Knee injury and Osteoarthritis Outcome Score Short Form), and VR-12 (Veterans RAND 12 Item Health Survey) Scale.

ELIGIBILITY:
Inclusion Criteria:

* adult (male and female) subjects aged 18 to 75,
* English speaking,
* are scheduled for primary total knee arthroplasty with planned spinal anesthesia with saphenous peripheral nerve block at the adductor canal.

Exclusion Criteria:

* general anesthesia,
* hepatic & renal failure,
* history of diabetic peripheral neuropathic pain,
* chronic opioid use,
* concurrent use of antidepressants, triptans, and/or linezolid,
* allergy to the study medications,
* prior knee surgery,
* BMI > 40,
* bleeding disorders,
* history of recent falls,
* concurrent benzodiazepine use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Cumulative 24 hour total opioid consumption | 24 hours
  morphine miligram equivalent

SECONDARY OUTCOMES:
Pain numeric rating scale at 24 hours post operatively | 24 hours
  Pain Scores will be measured on the Numerical Rating Scale (NRS), the score ranges from 0-10, zero indicating no pain and 10 indicating the worst pain.
Pain severity and interference at 7 days post operatively | 7 days
  The Brief Pain Inventory (BPI) assesses the severity of pain and its impact on functioning.The BPI scale defines pain as follows:1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Pain severity and interference at 3 months post operatively | 3 months
  The Brief Pain Inventory (BPI) assesses the severity of pain and its impact on functioning.The BPI scale defines pain as follows:1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Functionality at 7 days postoperatively | 7 days
  Knee injury and osteoarthritis outcome score short form: Patient-Reported Outcomes Measurement Information System (PROMIS), item health survey. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The average Score is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Functionality at 7 days postoperatively | 7 days
  Knee injury and osteoarthritis outcome score short form, veterans RAND 12 (VR12) item health survey. The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Therefore, each increment of 10 points above or below 50 corresponds to one standard deviation away from the population average.
Functionality at 3 months postoperatively | 3 months
  Knee injury and osteoarthritis outcome score short form: Patient-Reported Outcomes Measurement Information System (PROMIS), item health survey. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The average Score is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Functionality at 3 months postoperatively | 3 months
  Knee injury and osteoarthritis outcome score short form, veterans RAND 12 (VR12) item health survey. The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Therefore, each increment of 10 points above or below 50 corresponds to one standard deviation away from the population average.
Opioid consumption at 7 days postoperatively | 7 days
  morphine miligram equivalent
Opioid consumption at 3 months postoperatively | 3 months
  morphine miligram equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Behrends, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share our raw clinical data with other researchers.
Supporting Information: Study Protocol
Time Frame: For the entire study period
Access Criteria: Non-profit and research purpose.